CLINICAL TRIAL: NCT00340223
Title: Comparison of HIV-1 Epitopes That May be Recognized by HLA-B*3501 (PY) and -B*3503 (Px) Early After Seroconversion and After Development of AIDS
Brief Title: HLA-B35 Alleles and AIDS
Status: Withdrawn | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905237; 05-C-N237
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: HIV-1; AIDS
Keywords: Immunity; Mutations; Viral Selection; Disease Progression; RNA
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Disease Progression

SUMMARY:
This study will identify variations in the genome of the human immunodeficiency virus (HIV) early after infection and following the development of AIDS. It will analyze genetic material and clinical data from HIV-positive individuals to assess differences in viral epitopes between patients with two different gene alleles (alternative forms of a gene)-B*3501 and B*3503. (An epitope is a molecular region on the surface of an antigen capable of eliciting an immune response and of combining with the specific antibody produced by such a response.)

HIV disease in people with the B*3503 allele progresses significantly faster than it does in people with the B*3501 allele. This study might provide information that is potentially useful in developing a successful HIV vaccine.

Blood samples and clinical data for analysis will be obtained from the Johns Hopkins Bloomberg School of Public Health; the University of Pittsburgh; the John H. Stroger, Jr. Hospital of Cook County; the Howard Brown Health Center; Northwestern University; and the University of California at Los Angeles.

DETAILED DESCRIPTION:
The purpose of this study is to identify variations in the genome of HIV early after infection and following the development of AIDS to determine the location of escape mutations that might provide information about potential B*35 epitopes. These data will be useful in explaining the difference in disease progression between individuals possessing B*35 Px alleles and those with B*35 PY alleles. We have previously shown that individuals with B*35 Px alleles progress at a significantly faster rate compared to those with B*35 PY alleles. This study might provide information which is potentially useful in the development of a successful HIV vaccine.

ELIGIBILITY:
* INCLUSION AND EXCLUSION CRITERIA:

Sera and relevant clinical data from properly consented HIV positive seroconverters will be provided to the LGD for analysis. No available subjects will be excluded to maximize power. We will request an accrual ceiling of 100 participants.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-09; Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of California, Los Angeles, Los Angeles, California
  - Northwestern University, Chicago, Illinois
  - Howard Brown Health Center, Chicago, Illinois
  - John H. Stroger, Jr. Hospital of Cook County, Chicago, Illinois
  - John Hopkins Bloomberg School of Public Health, Baltimore, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - University of Pittsburgh, Pittsburgh, Pennsylvania

REFERENCES:
- [Background] Kiepiela P, Leslie AJ, Honeyborne I, Ramduth D, Thobakgale C, Chetty S, Rathnavalu P, Moore C, Pfafferott KJ, Hilton L, Zimbwa P, Moore S, Allen T, Brander C, Addo MM, Altfeld M, James I, Mallal S, Bunce M, Barber LD, Szinger J, Day C, Klenerman P, Mullins J, Korber B, Coovadia HM, Walker BD, Goulder PJ. Dominant influence of HLA-B in mediating the potential co-evolution of HIV and HLA. Nature. 2004 Dec 9;432(7018):769-75. doi: 10.1038/nature03113. PMID 15592417